CLINICAL TRIAL: NCT01116037
Title: ATS 3f(r) Aortic Bioprosthesis Model 1000 Post Approval Study
Acronym: PAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to end study due to limited enrollment and study population
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2008 Rev. D
Record Dates: First submitted 2010-04-08; First posted 2010-05-04 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Heart Valve Diseases
Keywords: Diseased Heart Valve, Replacement, Aortic, Stentless
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATS 3f Aortic Bioprosthesis (Other): ATS 3f Aortic Bioprosthesis, Model 1000 (equine pericardial bioprosthesis)
  Interventions: Device: ATS 3f Aortic Bioprosthesis

INTERVENTIONS:
Device: ATS 3f Aortic Bioprosthesis — Equine Pericardial Bioprosthesis for replacement of diseased valve

SUMMARY:
The purpose of this clinical study is to determine if there is an increased incidence and rate of aortic regurgitation in younger (</= 70 years of age) patients implanted with the Model 1000 and undergoing isolated aortic valve replacement of his/her native aortic valve, or replacement of a failed prosthesis.

DETAILED DESCRIPTION:
A multi-center non-randomized trial designed to obtain 606 patient years. Each enrolled patient will be followed for a minimum of six (6) years. Preoperative, discharge or 30 days (whichever comes last), 3-6 month, and annual follow-up data are required.

ELIGIBILITY:
Inclusion Criteria:

* Patient is </= 70 years of age and requires isolated aortic valve replacement with or without concomitant procedures such as coronary artery bypass or another valve reconstruction. (The three remaining valves must be of native tissue).
* Patient is sufficiently ill to warrant replacement of his/her diseased natural or prosthetic valve (excluding the ATS 3f Aortic Bioprosthesis, Model 1000 bioprosthesis), based on standard cardiovascular diagnostic workups.
* Patient is in satisfactory condition, based on the physical exam and Investigator's experience, to be an average or better operative risk, (i.e., likely to survive three years postoperatively).
* Patient is geographically stable and willing to return to the implant center for follow-up visits.
* Patient has been adequately informed and consents to his/her participation in the clinical study, and of what will be required of him/her, in order to comply with the protocol.

Exclusion Criteria:

* Patient is older than seventy (70) years of age.
* Patient has a non-cardiac major or progressive disease, which in the Investigator's experience produces an unacceptable increased risk to the patient, or results in a life expectancy of less than 3 years.
* Patient is an intravenous drug and/or alcohol abuser.
* Female patient is pregnant (urine HCG test result positive), or lactating.
* Patient presents with active endocarditis.
* Patient presents with congenital bicuspid aortic anatomy.
* This patient presents with abnormal aortic root geometry.
* Patient has chronic renal failure or is on renal dialysis.
* Patient has a previously implanted prosthetic valve that is not being replaced by a study valve.
* Patient requires mitral, tricuspid or pulmonic valve replacement.
* Patient presents with dilatation of the ascending aorta, Marfan Syndrome, Ehlers-Danlos syndrome, cystic medial degeneration, or other condition causing the ascending aorta to be irregular in geometry or physiology as seen via preoperative imaging.
* Patient is participating in concomitant research studies of investigational products.
* Patient will not agree to return to the implant center for the required number of follow-up visits or is geographically unavailable for follow-up.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Palmer, Study Director — Medtronic
Locations (6):
- United States (5):
  - Cardiac Surgery Clinical Research Center, Inc., Oak Lawn, Illinois
  - Columbia University, New York, New York
  - Univ of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Main Line Health Heart Center, Wynnewood, Pennsylvania
  - Baylor University, Dallas, Texas
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- See also: Medtronic Corporate Website — http://www.medtronic.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATS 3f Aortic Bioprosthesis
Started | 26
Completed | 1
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | ATS 3f Aortic Bioprosthesis
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Region of Enrollment [Count of Participants; unit: Participants] — Recruiting sites included 4 in the US (n=9) and 1 in Canada (n=17)
  Participants
    Canada | 17
    United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Goal is to Assess the Freedom From Clinically Significant (Moderate or Greater) Aortic Regurgitation for the Patients Implanted With 3f Aortic Bioprothesis, Model 1000
Description: Freedom from clinically significant (moderate or greater) aortic regurgitation will be determined through echocardiography and compared against the freedom from regurgitation event rates from the previous IDE study, G010284 used for PMA approval.
Time Frame: Six Years
Measure: Count of Participants; unit: Participants
Arm/Group | ATS 3f Aortic Bioprosthesis
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Safety Analysis Will be Based on the Occurence of Cardiovascular Complications.
Description: Safety Analysis will be based on the the number of participants with cardiovascular complications.
Time Frame: Six Years
Measure: Number; unit: participants
Arm/Group | ATS 3f Aortic Bioprosthesis
Number analyzed (Participants) | 26
participants | 11

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | ATS 3f Aortic Bioprosthesis
Serious Adverse Events (participants affected / at risk) | 8/26
Other Adverse Events (participants affected / at risk) | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATS 3f Aortic Bioprosthesis (N=26)
Cardiovascular Complications (Cardiac disorders) | 8 (10)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATS 3f Aortic Bioprosthesis (N=26)
Valve Dysfunction (Cardiac disorders) | 3 (3)
Vascular Complication (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No